CLINICAL TRIAL: NCT02283541
Title: Investigating the Relationship Between Gait, Depression, and Mind-body Therapy in Seniors
Brief Title: Gait, Depression, and Mind-body Therapy in Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Akshya Vasudev, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSREB 105915
Record Dates: First submitted 2014-10-29; First posted 2014-11-05 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Major Depressive Disorder
Keywords: Gait; late life depression; mind-body therapies
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASTM (Experimental): Participants in Automatic self-transcending meditation (ASTM) arm will complete a 12 week meditation training program in addition to their existing treatment plan. This involves participating in 120-minute sessions on each of four consecutive days of the first week. Participants will individually be given a mantra on day one, and then be instructed in use of the mantra according to specific criteria over the four session program. This will be followed by weekly 60-minute follow up sessions for the 11 subsequent weeks. In addition, participants will be asked to practice ASTM at home for 20 minutes twice daily over the study period. Assessments of depression severity will be completed at specific times over the 12 week training period: at Weeks 0, 4, 8 and 12.
  Interventions: Behavioral: Automatic self-transcending meditation
- TAU (No Intervention): Participants in TAU arm will continue with their existing treatment schedule as usual. Assessments of depression severity will be completed at specific times over the 12 week training period: at Weeks 0, 4, 8 and 12. However, no assessments will be done or information collected on the TAU arm from week 12 onwards. After week 12, TAU arm participants will be offered the opportunity to learn ASTM and attend follow up meditation.

INTERVENTIONS:
Behavioral: Automatic self-transcending meditation — ASTM is a category of meditation that helps quiet the mind and induce physiological and mental relaxation while the eyes are shut. It utilizes relaxed attention to a specific sound value (mantra) according to specific criteria, in order to draw attention inward.
  Other Names: ASTM
  Arms: ASTM

SUMMARY:
Falls are the leading cause of injury---related hospitalization and death in the elderly. As such, fear of falling (FOF) is common among senior populations and often leads to activity avoidance, social isolation, and reduced physical and mental health. Risk of falls is particularly concerning for individuals suffering from late life depression (LLD) as both depression and antidepressant treatment have been shown to be linked to gait impairments, a strong predictor of fall risk. Currently, our team is conducting a study to examine the effects of a non---pharmacological mind---body therapy commonly known as automatic self---transcending meditation (ASTM) on autonomic and mood---related symptoms of LLD. This study provides a timely opportunity to explore the intricate relationship between gait disturbances and depression severity, as well as the potential benefits of ASTM intervention on gait and FOF in seniors. Using a GAITRite® portable walkway, measures of stride length and gait velocity will be obtained for seniors in the ASTM and control study arms every four weeks for the duration of the ASTM program. The aim of this study is to answer the following research questions: are gait impairments and depression severity correlated, and does ASTM training have any effect on gait and FOF? The results of this study could not only provide insight into the physical manifestations of depression but if ASTM training is found to improve gait and reduce FOF then there is potential to use this mind---body meditation technique as an adjunct therapy to reduce fall risk in seniors with LLD. Furthermore, future research could expand upon these findings to examine the benefits of ASTM on gait impairments secondary to other psychiatric illnesses.

DETAILED DESCRIPTION:
Falls are the leading cause of injury---related death in senior populations (i.e. 65 years of age and older)

1. ; approximately 30% of community---dwelling seniors suffer a fall at least once per year, with this proportion increasing with age
2. . In Canada, 40% of falls by seniors result in hip fractures which oftentimes leads to only partial recovery
3. , therefore it is not uncommon for older adults to report a fear of falling (FOF). FOF is particularly common in community---dwelling older females and those who have previously experienced a fall [4,5]. In some individuals, FOF actually leads to activity avoidance

[5]. Moreover, seniors who have suffered a fall report reductions in their quality of life [6]. A systematic review by Scheffer et al. [4] has identified the major outcomes of FOF to be reductions in physical and mental health, quality of life and an increased risk of fall. Older adults suffering symptoms of depression are also more likely to have a severe FOF, leading to activity restriction in this group [7, 8]. As such, minimizing the risk of falls in older populations has important implications for the physical and mental wellbeing of individuals in this cohort. Among the risk factors that increase the likelihood of seniors suffering a fall are gait impairments [9] and depression [10---12]. Indeed, measures of gait can be used to predict future falls [13] while increases in depressive symptoms are associated with increases in fall rate [10]. An association has been established between depression and gait deficits, even when confounding variables such as socio---demographic and overall health status are controlled; specifically, depression is associated with reductions in various gait parameters including gait velocity, stride length and swing time variability [14, 15]. At present, antidepressants are the first line of treatment for depression, however in seniors the response rate to an antidepressant trial of adequate dose and duration is often inadequate and can be as low as 30--- 40% [16]. In addition, antidepressant use is often associated with a number of adverse events including increased fall risk [11] and impairments in gait [17, 18]. For example, in healthy seniors, a single dose of amitriptyline led to gait impairments when subjects were required to walk in the presence of obstructions [17]. Therefore the relationship between depression, gait, and fall risk is further complicated by standard pharmacological treatment practices for this population. In recent years, various non---pharmacological interventions have been embraced by patients with late life depression (LLD). Loosely defined as mind---body therapies, these include biofeedback, energy healing, meditation, guided imagery, and yoga [19, 20]. Amongst these practices, meditation therapy may be of particular benefit for older adults with gait impairments and LLD; meditation is non---invasive, easy to learn, has negligible side effects, can be practiced from anywhere and has been shown to have multi---organ benefits [see 21 for a review]. Whilst relatively few studies have examined the effects of meditation on gait, a study of mindfulness---based cognitive therapy (MBCT) found the therapy normalized gait patterns in adults with a history of depression [22]. Additionally, a particular type of meditation, referred to as automatic self---transcending meditation (ASTM) has been shown to reduce symptoms of depression [23]. Currently, our research team is commencing the data collection phase of an REB approved study that has received funding by the Academic Medical Organization of Southwestern Ontario (AMOSO) Innovation Fund. This study is a single blind longitudinal naturalistic randomized control trial targeting individuals with late---life depression, and will examine the effects of ASTM on autonomic and mood---related symptoms of depression. In the framework of the ASTM study there is an opportunity to more closely examine the relationship between gait and depression in elderly populations, as well as the potential benefits of this mind---body therapy on gait and FOF. We are kindly requesting funding from the Department of Psychiatry to carry out this investigation. Specifically, we aim to assess gait parameters such as stride length and gait velocity, which have been shown to be affected by depression [14, 15], in LLD patients receiving ASTM training in addition to their current treatment schedules (ASTM group) as well as those that continue with their treatment as usual (TAU group). A thorough literature and clinical trial registry search reveals that no one has previously, or is currently, examining the effects of ASTM training on parameters of gait in LLD patients.

ELIGIBILITY:
Inclusion Criteria:

* participants must be at least 65 years of age
* have a diagnosis of mild to moderate MDD with a 17 item Hamilton Depression Rating Scale (HAMD-17) score of 8 to 22
* be of good general physical health
* have sufficient hearing to be able to follow verbal instructions
* be able to sit without physical discomfort for 45 minutes and be able to attend 4 initial ASTM training sessions. They must also agree to home practice of ASTM and to attend 75% of weekly follow-up sessions.

Exclusion Criteria:

* potential participants must also be free of any physical impairments that would cause discomfort/stress when walking or affect our ability to obtain a representative measure of gait including injuries of the spinal cord, leg or foot, muscular dystrophy, multiple sclerosis, spinal stenosis, scoliosis, spondylolithesis, and severe osteoarthritis or rheumatoid arthritis of the spine.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean stride length at 4 weeks | Week 4
  Participants will be asked to complete three walks at their normal pace, beginning and ending 1m from the walkway to account for acceleration and deceleration. Baseline measures of mean stride length and gait velocity will be obtained. A mean gait velocity less than 100cm/s will be classified as a gait disorder
Change from baseline in mean stride length at 8 weeks | Week 8
  As above
Change from baseline in mean stride length at 12 weeks | Week 12
  As above
Change from baseline in mean stride length at 24 weeks | Week 24
  As above

SECONDARY OUTCOMES:
Change from baseline in gait velocity at 4 weeks | Week 4
  As above
Change from baseline in gait velocity at 8 weeks | Week 8
  As above
Change from baseline in gait velocity at 12 weeks | Week 12
  As above
Change from baseline in gait velocity at 24 weeks | Week 24
  As above

CONTACTS AND LOCATIONS:
Overall Officials: Akshya Vasudev, MBBS, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] 1. Liu E, Vasudev A. Primary Care Companion CNS Disord. 2014;16(3). DOI: 10.4008/PCC.14/0. 2. Gupta A, Bevan R, Vasudev A. Clinical Governance. 2014;19(2):83. 3. Vasudev A, et al. Current Reviews in Psychiatry. Forthcoming 2014. 4. Maldeniya P, Vasudev A. Case Reports in Psychiatry, 2013;432568. 5. Vasudev A. 2013. Manic syndromes in old age; p581. 6. Vasudev A, et al. Cochrane Database of Systematic Reviews. 2013;4:CD010495. 7. Vasudev K, Vasudev A. Commentary on Mitchell AJ, et al. Br J Psychiatry, 2012 Dec;201:435. Evidence Based Mental Health. 2013;16(2):58. DOI: 10.1136/eb-2012. 8. Colloby SJ, Firbank MJ, He J, Thomas AJ, Vasudev A, et al. British Journal of Psychiatry. 2012;200:150. 9. Colloby SJ, Firbank MJ, Vasudev A, et al. Journal of Affective Disorders. 2012;133(1-2):158. 10. Vasudev A, et al. Cochrane Database of Systematic Reviews. 2012;12:CD004694. 11. Vasudev A, et al. American Journal of Geriatric Psychiatry. 2012;20(8):691. 12. Colloby SJ, Vasudev A, et al. British Journal of Psychiatry. 2011;199(5):404. 13. Colloby SJ, Firbank MJ, Thomas AJ, Vasudev A, et al. Journal of Affective Disorders. 2011;135(1-3):216. 14. Vasudev A, et al. Cochrane Database of Systematic Reviews. 011;12:CD004857. 15. Vasudev A, et al. Depression in diabetes of the older person. United Kingdom: Springer; 2011.